CLINICAL TRIAL: NCT01028157
Title: STARS: Sistas Talking About Real Solutions
Brief Title: S.T.A.R.S.: Sistas Talking About Real Solutions
Acronym: STARS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gina M Wingood, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0524-2002; 5R01MH062717 (NIH)
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: HIV Prevention
Keywords: HIV; risk reduction; behavioral intervention
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Numbers Needed To Treat; Health Status; Nutritional Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Health Control (Placebo Comparator)
  Interventions: Behavioral: General Health & Nutrition
- HIV Risk Reduction & Relapse Prevention (Experimental)
  Interventions: Behavioral: STARS: Sistas Talking About Real Solutions

INTERVENTIONS:
Behavioral: STARS: Sistas Talking About Real Solutions — The intervention consisted of 2, 4-hour workshops. The first workshop focused on enhancing ethnic/gender pride, self-esteem, realizing values/setting goals, healthy/unhealthy relationships, partner violence, HIV/STD knowledge, heightening awareness of HIV susceptibility, safer-sex options/skills. The second workshop covered realistic choices in sexual decision making, consistent/proper condom use, setting limits/boundaries, communication styles, and condom skills negotiation. Participants received 3-hour booster sessions at 6- and 9-months to reinforce materials from the initial intervention. Bi-monthly phone calls and quarterly mailings were used to reinforce workshop material and facilitate retention.
  Other Names: Risk reduction; safer sex options
  Arms: HIV Risk Reduction & Relapse Prevention
Behavioral: General Health & Nutrition — Participants in this condition received a 2 hour group session which consisted of general health information and women's health brochures facilitated by a trained health educator. The control group received bi-monthly phone calls and quarterly mailings for retention purposes only, with no intervention material provided.
  Other Names: Placebo; Control; Health Control
  Arms: General Health Control

SUMMARY:
STARS: Sistas Talking About Real Solutions is a health education intervention for African-American women, ages 18-29 aimed at reducing their risk for HIV. A total of 855 subjects were recruited from three Kaiser Permanente Medical Centers. Members were randomly selected from the membership database and sent a letter via mail introducing them to the project and inviting them to participate. Letters were followed up with a phone call and potential participants were screened for eligibility. To be able to participate, participants had to be African-American, female, between the ages of 18-29, single, and have at least one act of unprotected sexual intercourse within the last 6 months. Members who were eligible and willing to participate completed a 1-hour baseline assessment survey; STD testing for Chlamydia, gonorrhea, trichomoniasis, and HPV; a vaginal swab that was used to determine if they had unprotected sex. They were then randomized into one of two study conditions: (1) a 2-session HIV risk-reduction condition with a safer sex relapse prevention component (2) a 1-session control condition in which participants receive general women's health information and brochures. Participants received a booster session at 6 and 9 months to reinforce intervention materials. Participants completed an assessment survey and received STD testing at 6 and 12 months. The primary aim of this project is to evaluate the efficacy of the HIV risk-reduction/safer sex relapse prevention condition relative to the health and nutritional control group in reducing HIV-associated sexual behaviors and incident STDs over a 12-month follow-up period is to implement.

DETAILED DESCRIPTION:
The primary aims of the study are: 1) to evaluate the efficacy of the HIV risk-reduction, safer sex relapse prevention condition relative to the general health and nutrition control condition in reducing HIV-associated sexual behaviors and incident STDs over a 12-month follow-up period; 2) to evaluate the efficacy of the HIV risk-reduction, safer sex relapse prevention condition relative to the general health and nutrition control condition in enhancing theoretically-derived mediators of HIV-preventive behaviors.

The study began recruitment into the main trial in October, 2002. By the close of the recruitment window in March 2006, 855 African American women had been randomized to either of the study conditions. The study participants were eligible if they were: (a) unmarried, (b) African American women, (c) ages 18-29, (d) not pregnant, (e) reported at least one act of unprotected sexual intercourse within the last 6 months and, (f) were members of one of the three Kaiser Permanente HMO study sites. The three medical facilities included the Cascade Kaiser Permanente Center, the Southwood Kaiser Permanente Center and, the Panola Kaiser Permanente Center. While there are other Kaiser Permanente Medical facilities in Atlanta, these sites were selected because of the high prevalence of African-American women.

Once recruited via a random selection process, participants returned to a Kaiser Medical Center on a specified Saturday morning for their baseline visit. At the baseline visit participants were: (1) provided a brief overview of the STARS study; (2) provided written informed consent; (3) asked to complete a one hour ACASI survey; (4) asked to provide self-obtained vaginal swab specimen that were assessed for four STDs (Chlamydia, gonorrhea, trichomonas, and human papilloma virus) and a new PCR procedure to detect the presence of sperm in vaginal specimen and; (5) randomized to one of the two study conditions using concealment of allocation techniques to minimize assignment bias.

The ACASI is guided by the Theory of Gender and Power and Social Cognitive Theory. The interview has sections on sociodemographics, sexual history, alcohol and drug use, attitudes and outcome expectations related to abstinence and condom use, peer norms, and stress and coping. The administration of the ACASI interview was enhanced by the inclusion of a 60-day calendar that participants complete prior to the interview. This allows a more realistic time frame to reference interview questions and time for the participant to recall and document behavior before beginning the interview. Upon completion of the full assessment, participants provided swabs for STI specimens. All participants with a positive test result were offered free directly observed therapy (DOT) at their participating medical center.

Participants were randomized to one of two study conditions: (1) an HIV safer sex risk-reduction condition with a relapse prevention component and; (2) a general health and nutrition control condition. the HIV safer sex risk-reduction condition consisted of two 4-hour safer sex workshops; the two workshops were guided by the Theory of Gender and Power and Social Cognitive Theory and; held on consecutive Saturdays at the participating medical centers. The sessions were implemented by a team of African American female health educators and had on average of 6 - 8 participants per session. The two study conditions are outlined below:

The HIV safer sex risk-reduction condition with a relapse prevention component: Participants in this condition received the two 4-hour safer sex workshops. The first workshop focused on enhancing ethnic and gender pride, self-esteem, realizing values and setting goals, healthy vs. unhealthy relationships, HIV/STD knowledge, heightening awareness of HIV susceptibility, safer-sex options. The second workshop offered realistic choices in sexual decision making, covering topics including abstinence, masturbation, oral, vaginal, and anal sex. The risk and benefits related to each safer-sex option were examined. Participants also received instruction on safer-sex skills corresponding to each option. Consistent and proper condom use was also discussed and demonstrated with a module on condom skills. This module included activities demonstrating the increased difficulty of proper condom use when under the influence of substances such and drugs and alcohol. Modules on setting limits and boundaries, communication styles, and condom skills negotiation were also a part of this workshop. In addition, an activity was included on indications and ways to deal with partner violence. Workshop II included several role-play scenarios demonstrating how to handle excuses related to safer-sex options and also exhibiting realistic situations that women may face in their sexual relationships. Participants in this condition received 3-hour booster sessions at 6- and 9-months to reinforce materials from the initial intervention. The 6-month booster session included modules that reinforced concepts such as gender and ethnic pride, self-esteem, communicating safer-sex options, assertive communication skills, difficulties communicating with long-term partners, and standing by one's safer-sex decisions. Again, role plays and interactive activities facilitated participants' ability to explore and examine challenges they experienced related to these topics. In a similar fashion, the 9-month booster session reinforced positive safer-sex messages, exploration of past unsafe sexual experiences, mastering safer sex techniques, identifying and making wise decisions about healthy and unhealthy partner characteristics, creative options for safer sex, gender and ethnic pride, and empowerment to make and maintain healthy choices. Bi-monthly phone calls and quarterly mailings were used to reinforce workshop material and facilitate retention.

The control condition: Participants in this condition received a 2 hour group session which consisted of general health information and women's health brochures facilitated by a trained health educator. The control group received bi-monthly phone calls and quarterly mailings for retention purposes only, with no intervention material provided.

Participants in all study conditions received a group introduction including group guidelines, definition of a 'STARS Sista', the STARS motto, pact and group contract.

Follow-up visits: At the 6-month follow-up visit all participants completed the 6-month ACASI to assess potential behavior change and change in the study mediators; and provided specimens for Chlamydia, gonorrhea and trichomoniasis; and provided a specimen for the PCR procedure to detect the presence of sperm in a vaginal sample.

At the 12-month follow-up visit participants completed the 12-month ACASI to assess potential behavior change and change in the study mediators; provided specimens for Chlamydia, gonorrhea and trichomoniasis and HPV (if they did not test positive for HPV at baseline); and provided a specimen for the PCR procedure to detect the presence of sperm in a vaginal sample.

ELIGIBILITY:
Inclusion Criteria:

* African American
* female
* Age 18-29
* unmarried
* engaged in at least one act of unprotected sexual intercourse within the last 6 months
* were members of one of the three Kaiser Permanente HMO study sites

Exclusion Criteria:

* pregnant or trying to get pregnant
* young adults who have a condition that precludes participation (i.e. schizophrenia, severe learning disability, or undergoing chemotherapy)

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 855 (Actual)
Dates: Start 2002-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of a HIV risk-reduction condition relative to general health control condition in reducing HIV-associated sexual behaviors and incident STDs. | 12 months

SECONDARY OUTCOMES:
To evaluate the efficacy of a HIV risk-reduction condition relative to general health control condition in enhancing theoretically-derived mediators of HIV-preventive behaviors. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gina M Wingood, ScD, MPH, Principal Investigator — Emory University; LaShun R Robinson, PhD, Study Director — Emory University; Ralph DiClemente, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Rollins School of Public Health, Atlanta, Georgia, United States